CLINICAL TRIAL: NCT00867360
Title: Hypothalamic-Pituitary-Adrenal (HPA)/Dopamine Axis in Psychotic Depression
Brief Title: Treatment of Psychotic Major Depression With Mifepristone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alan Schatzberg, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-02262009-1838
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Affective Disorders, Psychotic; Depressive Disorder
MeSH Terms: conditions — Affective Disorders, Psychotic; Depressive Disorder | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Experimental): Receive mifepristone for 8 days
  Interventions: Drug: Mifepristone (RU-486)
- Placebo (Placebo Comparator): Receive placebo rather than mifepristone
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone (RU-486)
  Arms: Mifepristone
Drug: Placebo — Placebo medication
  Arms: Placebo

SUMMARY:
The purpose of this research study is to see how certain hormones cause changes in mood and thinking in some depressed patients and to determine the effectiveness of mifepristone in treating some forms of depression.

This study is conducted in conjunction with an observational study "Clinical and Biological Characteristics of Psychotic Depression".

DETAILED DESCRIPTION:
Eligibility Procedures: Before entering the study and prior to any other procedures, you will be asked to read and sign this consent form. To determine if you are eligible for our study, you will then have a general medical (including menstrual cycle history on female patients) and psychiatric history taken, a physical examination, your vital signs (blood pressure, pulse), height, weight and waist/hip ratio will be measured, as well as various psychiatric evaluations will be conducted.

You will be randomly (by chance) assigned to receive mifepristone or placebo (an inactive substance). Half of the participants in this research study will receive placebo, and half will receive mifepristone. Neither you nor your study doctor will know which of the two you are receiving. Treatment will begin in the morning of Treatment Day 1 and conclude on Treatment Day 8 for a total treatment period of 8 days. You will take the medication once a day in the morning. The dose was originally 600 mg but was changed to 1200 mg per day after the 4th patient. You will not be able to take any new medications (other than the study drug) or make changes to your current medications while participating in this part of the study unless ordered by the study physician.

On treatment Day 1, you will come to our office for an interview and we will evaluate your mood and other psychiatric symptoms. Additionally, we will take your vital signs and draw blood to administer clinical laboratory tests. You will meet with the study physician and will then be given 4-days of medication to take home with you and self-administer each morning.

On Treatment Day 4, you will come back to our office. We will evaluate your mood, take your vital signs and you will meet with the study physician. It is important that you discuss with your study physician or the research study staff all unpleasant or unusual symptoms that you may experience. Any positive effects that are experienced should be discussed as well. You will be given an additional 4-days of medication to take home with you to self-administer each morning.

On Treatment Day 8, we will re-evaluate your mood, take your vital signs and repeat the blood and urine lab tests. You will also meet with the study physician to discuss any side effects. If you are participating in the blood draw portion of this study, you will be admitted to the GCRC on this day for an overnight stay. At 2pm on Treatment Day 8, you will have an IV line inserted into one arm for hourly blood samples from 2pm, 4pm, then 6pm until 9am on Treatment Day 9. At 9am on treatment Day 9, 10 mls of blood will be taken for Mifepristone concentration. A total of 82mls (approximately 5.5 tablespoons) of blood will be drawn. You will be discharged from the GCRC following breakfast.

On Treatment Day 15, we will re-evaluate your mood and you will meet with the study physician to discuss any side effects.

On Treatment Day 22, you will be readmitted to the GCRC, where nurses will take your vitals signs and repeat the clinical laboratory tests. We will also reevaluate your mood, and you will meet with the study physician to discuss any side effects. If you have participated in portions or all of the baseline protocol (protocol # 13088) you will repeat neuropsychological, MRI and blood draw procedures accordingly. If you did not participate in the baseline protocol, you will be assessed for safety and discharged.

You will have another functional MRI (a picture taken of your brain using a magnet while you are administered a series of tasks). This MRI scan procedure will take approximately 1 hour. You will be given a series of neuropsychological tests to assess your memory and concentration. You will be asked to complete several questionnaires during your hospital stay. These questionnaires ask for your views about your personality, your childhood, your quality of life, your mood and a variety of aspects of your daily functioning. The questionnaires may be completed anytime during your overnight stay and will take about 2.5 hours to finish. On treatment Day 22, you will have an IV line inserted into one arm for hourly blood samples taken at 2pm, 4pm and then hourly from 6pm to 9am. A total of 72 ml's (approximately 5 tablespoons) of blood will be drawn.

At 2pm on Treatment Day 23, you will have another IV line placed in your arm to draw hourly blood samples used for the measure of ACTH and cortisol. These blood samples are taken in small amounts (approximately 1 teaspoon) and will be collected at 2pm and then on the hour, every hour, starting at 3pm and ending at 7pm, then every 30 minutes until 12pm. At 3pm, you will be given 0.5mg (five 0.1mg tablets) of Fludrocortisone. At 4pm, 10 mls of blood will be taken for Mifepristone concentration. Following the last blood draw at 12pm, a blood sample will be taken for clinical laboratory assessment to ensure your safety following Fludrocortisone administration. A total of 76ml's (approximately 5 tablespoons) of blood will be drawn. The IV line will then be removed and your vital signs will be assessed.

The following morning, the study physician will contact the experimental pharmacy and find out whether you have received placebo (no medication) or mifepristone. If you have been treated with mifepristone, this will mark the end of your study participation and the research coordinator will discuss follow-up assessments with you. The follow up assessments will be as follows: mood assessments will be performed via phone on weeks 1 and 2 and months 1, 3, 6, and 12 after completion of the study. These assessments will take a maximum of 1 hour to complete. The physician will also confirm your continued care and treatment with your primary treating psychiatrist. You will then be discharged from the GCRC and the hospital.

If you have been on the placebo, you will be offered an 8-day open-label trial of mifepristone.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for PMD (individuals with Psychotic Major Depression) are as follows:

1. DSM IV diagnosis of Major Depressive Disorder with psychotic features, Bipolar II Disorder with psychotic features in a major depressive episode.
2. 21-item HAM-D score greater than or equal to 21.
3. Thase Core Endogenomorphic Scale score greater than or equal to 6 on the items included in the 21-item HDRS.
4. Between 21 - 85 years of age.
5. Female patients of child bearing capacity with Psychotic Depression receiving treatment with mifepristone are required to use a double-barrier method of contraception or abstinence for the entire duration of the study as well as for thirty days after the last dose of Mifepristone is taken.
6. If currently taking antipsychotic, antidepressant, anticonvulsant, and/or mood-stabilizing medications, must be stable on the medication for at least one-week prior to entering the study.
7. Pre-existing (current) primary treating psychiatrist for subjects with psychotic features.
8. Any secondary diagnoses from the anxiety disorder spectrum is acceptable. Any secondary diagnoses from the anxiety disorder spectrum is acceptable. Primary pre-existing chronic Obsessive-Compulsive Disorder(OCD) will be an exclusion criteria. Exclusion Criteria:Exclusion criteria for PMDs are as follows:

1. ECT in the 6 months prior to the study. 2. Abuse of drugs or alcohol in the 6 months prior to study. 3. Unstable or untreated hypertension, cardiovascular disease. 4. If participating in the blood draw portion of the protocol, endocrine disorders are exclusionary. 5. Use of additional prescription medications, street drugs, or alcohol during the week before the study. 6. Previous mifepristone failure or non-response. 7. Any Axis II diagnosis or traits which would make participation in the study difficult. 8. Current pregnancy or lactation.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric B Kraemer, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone: Receive 1200 mg/ day of mifepristone for 8 days
  Mifepristone (RU-486)
Period: Overall Study
Arm/Group | Mifepristone | Placebo
Started | 4 | 6
Completed | 3 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.67 (13.1) | 40.00 (9.98) | 39.88 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Psychotic Symptoms Subscale (PSS) of the Brief Psychiatric Rating Scale (BPRS)
Description: The BRPS is a rating scale of various psychiatric symptoms. Each item is rated on a scale of 1 to 7, with 1 being not present. The PSS is the sum of 4 items from the BPRS, which indicates the level of positive psychotic symptoms.. Thus, the range for the PSS is 4 to 28, with higher scores indicating greater levels of positive psychotic symptoms.
  For ease of interpretation, the sum of the PSS then has 4 items subtracted so that a score of 0 (instead of 4) indicates that there are no psychotic symptoms. In doing this, the range for the PSS becomes 0 to 24), with larger values indicating more positive psychotic symptoms.
  The measure is the change score of PSS total day 1 less PSS total Day 9. 0 indicates no change, where as positive numbers indicate a decrease in psychotic symptoms.
Time Frame: baseline to day 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 3 | 5
units on a scale | .000 (2.6) | 1.00 (.625)

2. Primary Outcome: Change in Mean Cortisol Level
Description: The reported value is the difference in mean evening cortisol from baseline to Day 9 The mean evening cortisol is calculated from the hourly cortisol value taken from 1800 hrs to 0100 hrs for both time points. The outcome measure is the difference of mean evening cortisol from Day 9 less the mean evening cortrisol from baseline. Negative values indicate a reduction in cortisol levels at Day 9, whereas positive values indicate an increase in cortisol at Day 9. Serum cortisol levels are reported in ug/dL
Time Frame: Day 1 to Day 9 difference
Population: Change in cortisol from Day 1 to Day 9
Measure: Mean (Standard Deviation); unit: ug/dL
Groups:
- Mifepristone: Receive 600 or 1200 mg/ day of mifepristone for 8 days
  Mifepristone (RU-486)
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 3 | 5
ug/dL | -3.96 (2.4) | .285 (.95)

3. Secondary Outcome: % Change in Mean Evening Pre- and Post- Florinef Cortisol After Treatment With Either Mifepristone or Placebo
Description: Time 1 (baseline) = Difference in cortisol level from Day 1 (pre-florinef mean evening cortisol) at Baseline less Day 2 (post-florinef mean evening cortisol) at baseline
  Time 2 (post- mife or placebo treatment) = Difference in cortisol level from Day 22 (pre-florinef mean evening cortisol) and Day 23 (post-florinef mean evening cortisol level).
  All measurements were the percent change in mean cortisol level from 6 pm to 10 pm. Cortisol levels are expressed as ug/dL
  Percent change in cortisol decrease between Time 2 and Time 1 post florinef should be greater with mifepristone than placebo, reflecting enhanced mineralocorticoid receptor activity.
Time Frame: Day 23
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 2 | 5
percentage change | 14 (.13) | -.04 (.19)

ADVERSE EVENTS:
Time Frame: Adverse events were gather while participating in the protocol, approximately 2 weeks
Description: Information on other adverse events was not readily available at time of reporting.
Arm/Group | Mifepristone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=4) | Placebo (N=6)
Psychaitric decompensation requiring hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No